CLINICAL TRIAL: NCT01728454
Title: A Phase 2, Multi-Center, Three-Arm, Parallel Design, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of 6 and 12 mg Proellex® (Telapristone Acetate) Administered Orally in the Treatment of Premenopausal Women With Confirmed Symptomatic Endometriosis
Brief Title: Safety and Efficacy of Telapristone Acetate (Proellex®) in the Treatment of Pre-Menopausal Women With Confirmed, Symptomatic Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZPE-202
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Following the Stage 1 no treatment baseline assessment period, placebo matching capsules, orally, once daily for 18 weeks in Stage 2. Eligible participants had the option to receive 2 additional 16-week cycles of active treatment at 12 milligrams (mg)/day separated by an off-drug interval (ODI) in Stage 3.
  Interventions: Drug: Placebo
- Telapristone acetate 6 mg (Experimental): Following the Stage 1 no treatment baseline assessment period, telapristone acetate (Proellex®) 6 mg capsules, orally once daily for 18 weeks in Stage 2. Eligible participants had the option to receive 2 additional 16-week cycles of active treatment at 6 mg/day separated by an ODI in Stage 3.
  Interventions: Drug: Telapristone acetate
- Telapristone acetate 12 mg (Experimental): Following the Stage 1 no treatment baseline assessment period, telapristone acetate (Proellex®) 12 mg capsules, orally once daily for 18 weeks. Eligible participants had the option to receive 2 additional 16-week cycles of active treatment at 12 mg/day separated by an ODI in Stage 3.
  Interventions: Drug: Telapristone acetate

INTERVENTIONS:
Drug: Placebo — Placebo matching capsules, orally, once daily for 18 weeks.
  Arms: Placebo
Drug: Telapristone acetate — Telapristone acetate capsules, orally once daily for 18 weeks.
  Other Names: Proellex®
  Arms: Telapristone acetate 12 mg; Telapristone acetate 6 mg

SUMMARY:
The primary purpose of this study is to determine the safety and efficacy of two oral doses of telapristone acetate administered to premenopausal women with pelvic pain associated with endometriosis confirmed within the last seven years and using prescription analgesics for symptomatic pain.

DETAILED DESCRIPTION:
This study is a phase 2, 3-arm-study with an 18-week active dosing period and an option for participants to receive 2 additional 16-week cycles of active treatment at their randomized dose [6 mg or 12 mg/day]. Placebo participants who elect additional treatment will receive treatment at 12 mg/day. The treatment dose will remain double-blind. The study will be conducted in 3 stages. The first stage is a no treatment baseline assessment period. This stage will last as long as it takes to record at least one full menstrual cycle (ovulation until ovulation).

For stage 2, following the run-in stage, at Visit 3, 60 participants will be randomized into one of 3 arms in a 1-1-1 fashion. The start of dosing should commence as soon as possible after ovulation following the end of the previous menstrual event.

For stage 3, participants who are eligible to receive additional cycles of treatment and who elect to continue treatment will be scheduled within a week before the second expected menses (+/- 2 days), following the off-drug interval. Participants will receive 2 cycles of treatment separated by an off-drug interval (ODI), after which they will be followed until menses has returned.

ELIGIBILITY:
Inclusion Criteria:

* Adult females between 18 and 47 years of age using prescription analgesics for endometriosis pain and with a Biberoglu Behrman Symptom Severity Scale (BBSS) score ≥7 at screening (assessed over the previous 28 days).
* Endometriosis diagnosis must have been surgically confirmed within 7 years. A laparoscopic diagnosis is acceptable.
* Participants must have a history of at least 3 regular menstrual cycles in which symptoms of endometriosis occurred immediately prior to screening.
* Normal or abnormal but non-clinically significant transvaginal ultrasound.
* History of menstrual events occurring in regular cycles.
* Agreement not to attempt to become pregnant during the trial.
* Agreement to limit alcohol consumption to no more than 2 drinks per week and to avoid alcohol consumption within 48 hours before each visit.
* Ability to complete a daily electronic participant diary and study procedures in compliance with the protocol.
* Women of child-bearing potential must be willing to use double-barrier contraception during the study and for 30 days after discontinuation of study medication. Acceptable double-barrier methods are: male condom with spermicide; male condom with diaphragm; diaphragm containing spermicide plus additional intra-vaginal spermicide.
* Has a negative pregnancy test at the Screening and Baseline visits, and subsequent study visits.
* A Body Mass Index (BMI) between 18 and 39 inclusive.
* Is available for all treatment and follow-up visits.

Exclusion Criteria:

* Post-menopausal woman, defined as either; six (6) months or more (immediately prior to screening visit) without a menstrual period, or prior hysterectomy and/or oophorectomy.
* Pregnant or lactating or is attempting or expecting to become pregnant during the 6-7 month study period.
* Women with abnormally high liver enzymes or liver disease [alanine transaminase (ALT) or aspartate aminotransferase (AST) exceeding 2 x upper limit of normal (ULN) and total bilirubin exceeding 1.5 x ULN at screening and confirmed on repeat].
* Received an investigational drug in the 30 days prior to the screening for this study.
* History of polycystic ovary syndrome (PCOS).
* Concurrent use of any testosterone, androgen, anabolic steroids, dehydroepiandrosterone (DHEA) or hormonal products for at least 2 weeks prior to screening and during the study. Oral contraceptive use for control of endometriosis symptoms is acceptable for the first 28-days of the study.
* Use of Depo-Provera® in the preceding 6 months.
* Use of Gonadotrophin releasing hormone (GnRH) as (e.g. Lupron Depot) within 3 months of the first dose of study drug (Lupron Depot must have a wash-out period of 3 months after the period of duration of the Lupron dose).
* Has an intrauterine device (IUD) in place. Copper IUDs (non-hormone containing will be permitted).
* Presence of intramural fibroids that impact the endometrial stripe, submucosal fibroids (any size), or endometrial polyps. Subserosal and intramural fibroids with no impact on the endometrial stripe are acceptable.
* Presence of endometrioma(s).
* Present history or condition that causes non-endometriosis related dyspareunia (e.g. vulvar vestibulitis).
* Past or present history of thrombophlebitis or thromboembolic disorders.
* Known or suspected carcinoma of the breast or reproductive organs.
* History of abnormal electrocardiogram (ECG) that, in the opinion of the investigator, is clinically significant and will prevent the participant from completing the study, including a QTc (corrected QT interval) of greater than 450 milliseconds (ms).
* Cervical dysplasia classified as Atypical Squamous Cells of Undetermined Significance (ASCUS) associated with high-risk human papilloma virus (HPV) or Low/High Grade Squamous Intraepithelial Lesion (LGSIL or HGSIL).
* History of abnormal endometrial biopsy including the presence of Endometrial Intraepithelial Neoplasia (EIN).
* Recent history (within past 6 months) of alcoholism or drug abuse.
* Known active infection with Human Immunodeficiency Virus (HIV), Hepatitis A, B or C.
* Previous history of auto-immune disease and/or positive antinuclear antigen (ANA).
* Endometrial stripe ≥18 mm in thickness at Visit 1.
* Women currently taking cimetidine or spironolactone.
* Clinically significant abnormal findings on screening examination and laboratory assessments or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study.

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05-02 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (10):
- United States (10):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Jacksonville, Florida
  - Margate, Florida
  - Metairie, Louisiana
  - Summerville, South Carolina
  - Houston, Texas
  - Riverton, Utah
  - Salt Lake City, Utah
  - Richmond, Virginia

REFERENCES:
- [Derived] Rolla E. Endometriosis: advances and controversies in classification, pathogenesis, diagnosis, and treatment. F1000Res. 2019 Apr 23;8:F1000 Faculty Rev-529. doi: 10.12688/f1000research.14817.1. eCollection 2019. PMID 31069056
- See also: Sponsor corporate web page — http://reprosrx.com

RESULTS

PARTICIPANT FLOW:
Period: Stage 1 and 2
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Started | 17 | 20 | 23
Completed | 12 | 16 | 19
Not Completed | 5 | 4 | 4
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Non-compliance with Protocol | 0 | 0 | 1
Not completed — Moved to Active Drug/ Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrew due to Adverse Events/Toxicity | 2 | 3 | 3
Period: Stage 3
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Started | 6 (Eligible participants who opted to participate in Stage 3.) | 5 (Eligible participants who opted to participate in Stage 3.) | 11 (Eligible participants who opted to participate in Stage 3.)
Completed | 3 | 1 | 7
Not Completed | 3 | 4 | 4
Not completed — Reason Missing | 0 | 0 | 1
Not completed — Subject Required Other Treatment | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrew Consent | 1 | 0 | 1
Not completed — Non-compliance with Protocol | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Withdrew due to Adverse Events/Toxicity | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all study participants who were randomized, received study drug, and had some post-baseline safety data.
Groups:
- Placebo: Following the Stage 1 no treatment baseline assessment period, placebo matching capsules, orally, once daily for 18 weeks in Stage 2. Eligible participants had the option to receive 2 additional 16-week cycles of active treatment at 12 mg/day separated by an off-drug interval (ODI) in Stage 3.
- Total: Total of all reporting groups
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Total
Number analyzed (Participants) | 17 | 20 | 23 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (6.52) | 30.8 (5.93) | 30.1 (7.07) | 29.8 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 23 | 60
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 6 | 4 | 12
  White | 15 | 14 | 18 | 47
  Other | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 5 | 14
  Non-Hispanic or Non-Latino | 12 | 16 | 18 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Individual Biberoglu Behrman Symptom Severity Scale (BBSS) Score for Dysmenorrhea
Description: The BBSS scale defined dysmenorrhea according to the loss of work efficiency and need for bed rest. The dysmenorrhea was graded on a scale from 0 to 3 where, 0 = None; 1 = Mild (some loss in work efficiency); 2 = Moderate (in bed part of the day, occasional loss of work efficiency); 3 = Severe (in bed one or more days, incapacitation), with higher scores indicating more severe symptoms. Participants were provided with a daily diary to record information about participant-reported scores for endometriosis pain each day. Daily scores were standardized to a 28-day period for each interval (Baseline, On-drug Cycle 1 and Off-drug Cycle 1) calculated as the sum of scores in the interval divided by the number of the days in the interval multiplied by 28. A negative change from Baseline indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to the last day of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks) and at the end of Off-drug Cycle 1 (Off-drug Cycle 1 is 3 weeks following On-drug Cycle 1)
Population: Intent-to-Treat (ITT) population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: score on a scale per 28-day period
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
score on a scale per 28-day period
  Baseline | 12.6 (5.58) | 10.8 (6.90) | 11.1 (5.55)
  Change from Baseline to On-Drug Cycle 1 | -3.95 (5.936) | -8.46 (5.174) | -6.46 (10.668)
  Change from Baseline to Off-Drug Cycle 1: number analyzed (Participants) | 14 | 18 | 21
  Change from Baseline to Off-Drug Cycle 1 | -2.43 (7.852) | 1.36 (14.546) | -1.82 (9.054)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle 1; Test type: Superiority; p = 0.0360, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle 1; Test type: Superiority; p = 0.1087, Wilcoxon Rank- Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Off-Drug Cycle 1; Test type: Superiority; p = 0.2263, Wilcoxon Rank- Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Off-Drug Cycle 1; Test type: Superiority; p = 0.5375, Wilcoxon Rank- Sum Test

2. Primary Outcome: Change From Baseline in Individual BBSS Score for Dyspareunia
Description: The BBSS scale defined deep dyspareunia according to the limitation of sexual activity. The dyspareunia was graded on a scale from 0 to 3 where, 0= None (no discomfort); 1= Mild (tolerated discomfort); 2= Moderate (intercourse painful to the point of interruption); 3= Severe (intercourse avoided because of pain), with higher scores indicating more severe symptoms. Participants were provided with a daily diary to record information about participant-reported scores for endometriosis pain each day. Daily scores were standardized to a 28-day period for each interval (Baseline, On-drug Cycle 1 and Off-drug Cycle 1) calculated as the sum of scores in the interval divided by the number of the days in the interval multiplied by 28. A negative change from Baseline indicates improvement..
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: score on a scale per 28-day period
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
score on a scale per 28-day period
  Baseline: number analyzed (Participants) | 14 | 16 | 19
  Baseline | 41.2 (24.15) | 36.5 (24.43) | 39.8 (21.42)
  Change from Baseline to On-Drug Cycle 1: number analyzed (Participants) | 12 | 16 | 18
  Change from Baseline to On-Drug Cycle 1 | -21.50 (18.800) | -14.75 (19.749) | -9.83 (15.594)
  Change from Baseline to Off-Drug Cycle 1: number analyzed (Participants) | 12 | 16 | 18
  Change from Baseline to Off-Drug Cycle 1 | -21.50 (18.800) | -14.75 (19.749) | -9.83 (15.594)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle 1; Test type: Superiority; p = 0.1017, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle 1; Test type: Superiority; p = 0.1927, Wilcoxon Rank- Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Off-Drug Cycle 1; Test type: Superiority; p = 0.1017, Wilcoxon Rank- Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Off-Drug Cycle 1; Test type: Superiority; p = 0.1927, Wilcoxon Rank- Sum Test

3. Primary Outcome: Change From Baseline in Individual BBSS Score for Non-Menstrual Pelvic Pain
Description: The BBSS scale defined non-menstrual pelvic pain according to various degrees of discomfort and use of analgesics. The non-menstrual pelvic pain was graded on a scale from 0 to 3 where, 0= None (absence of pain); 1= Mild (occasional pelvic discomfort); 2= Moderate (noticeable discomfort for most of the cycle); 3= Severe (pain persisting during the cycle or requiring strong analgesics), with higher scores indicating more severe symptoms. Participants were provided with a daily diary to record information about participant-reported scores for endometriosis pain each day. Daily scores were standardized to a 28-day period for each interval (Baseline, On-drug Cycle 1 and Off-drug Cycle 1) calculated as the sum of scores in the interval divided by the number of the days in the interval multiplied by 28. A negative change from Baseline indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to the last day dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks) and to the end of Off-drug Cycle 1 (Off-drug Cycle 1 is 3 weeks following On-drug Cycle 1)
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: score on a scale per 28-day period
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
score on a scale per 28-day period
  Baseline | 34.3 (18.07) | 33.5 (17.85) | 32.7 (16.68)
  Change from Baseline to On-Drug Cycle 1 | -6.06 (11.132) | -10.01 (15.200) | -2.96 (15.782)
  Change from Baseline to Off-Drug Cycle 1: number analyzed (Participants) | 14 | 18 | 21
  Change from Baseline to Off-Drug Cycle 1 | -6.87 (12.034) | -13.09 (17.745) | -8.26 (13.608)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle 1; Test type: Superiority; p = 0.7508, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle 1; Test type: Superiority; p = 0.5507, Wilcoxon Rank- Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; Off-Drug Cycle 1; Test type: Superiority; p = 0.3993, Wilcoxon Rank- Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; Off-Drug Cycle 1; Test type: Superiority; p = 0.5821, Wilcoxon Rank- Sum Test

4. Secondary Outcome: Change From Baseline in Prescription Analgesics Usage
Description: An analgesic was any member of the group of drugs used to achieve analgesia, relief from pain. Prescription analgesics are analgesics prescribed by the physician. Participants were provided with a daily diary to record the number of pills of non-narcotic prescription and narcotic analgesics taken for endometriosis-related pain symptoms each day. Daily number of pills were standardized to a 28-day period for each interval (Baseline and On-drug Cycle 1) calculated as the sum of pills in the interval divided by the number of the days in the interval multiplied by 28. A negative change from Baseline indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to the last day of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks)
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: pills per 28-day period
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
pills per 28-day period
  Baseline | 14.8 (18.13) | 14.9 (20.72) | 31.4 (52.55)
  Change from Baseline to On-Drug Cycle | -6.74 (14.897) | -7.20 (15.948) | -5.87 (27.753)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle; Test type: Superiority; p = 0.7507, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle; Test type: Superiority; p = 0.8919, Wilcoxon Rank- Sum Test

5. Secondary Outcome: Percentage Change From Baseline in Prescription Analgesics Usage
Description: An analgesic was any member of the group of drugs used to achieve analgesia, relief from pain. Prescription analgesics are analgesics prescribed by the physician. Participants were provided with a daily diary to record the number of pills of non-narcotic prescription and narcotic analgesics taken for endometriosis-related pain symptoms each day. Daily number of pills were standardized to a 28-day period for each interval (Baseline and last 28-days On-drug Cycle 1) calculated as the sum of pills in the interval divided by the number of the days in the interval multiplied by 28.The percent change from baseline in the analgesic usage was determined by subtracting the baseline analgesic usage from the analgesic usage during the last nominal 28 day menstrual cycle, divided by the baseline analgesic usage, and multiplied by 100%. A negative percent change from Baseline indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to last 28 days of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks)
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
percent change | -9.69 (71.980) | -21.63 (76.530) | -6.36 (174.210)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle; Test type: Superiority; p = 0.4780, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle; Test type: Superiority; p = 0.2354, Wilcoxon Rank- Sum Test

6. Secondary Outcome: Change From Baseline in Non-Prescription Analgesics Usage
Description: An analgesic was any member of the group of drugs used to achieve analgesia, relief from pain. Nonprescription analgesics are over-the-counter (OTC) analgesics. Participants were provided with a daily diary to record the number of pills of OTC drugs taken for endometriosis-related pain symptoms each day. Daily number of pills were standardized to a 28-day period for each interval (Baseline and On-drug Cycle 1) calculated as the sum of pills in the interval divided by the number of the days in the interval multiplied by 28. A negative change from Baseline indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to last day of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks)
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: pills per 28-day period
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
pills per 28-day period
  Baseline | 19.0 (29.05) | 15.4 (26.95) | 43.2 (98.60)
  Change from Baseline to On-Drug Cycle | 1.78 (21.426) | -12.79 (25.628) | -6.81 (25.615)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle; Test type: Superiority; p = 0.1140, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle; Test type: Superiority; p = 0.1636, Wilcoxon Rank- Sum Test

7. Secondary Outcome: Percentage Change From Baseline in Non-Prescription Analgesics Usage
Description: An analgesic was any member of the group of drugs used to achieve analgesia, relief from pain. Nonprescription analgesics are OTC analgesics. Participants were provided with a daily diary to record the number of pills of over the counter drugs taken for endometriosis-related pain symptoms each day. Daily number of pills were standardized to a 28-day period for each interval (Baseline and last 28-days On-drug Cycle 1) calculated as the sum of pills in the interval divided by the number of the days in the interval multiplied by 28. The percent change from baseline in the analgesic usage was determined by subtracting the baseline analgesic usage from the analgesic usage during the last nominal 28 day menstrual cycle, divided by the baseline analgesic usage, and multiplied by 100%. A negative percent change indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to last 28 days of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks)
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
percent change | 6.06 (62.237) | -22.80 (57.498) | -31.49 (60.114)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle; Test type: Superiority; p = 0.1140, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle; Test type: Superiority; p = 0.0733, Wilcoxon Rank- Sum Test

8. Secondary Outcome: Change From Baseline in Total Analgesics Usage
Description: An analgesic was any member of the group of drugs used to achieve analgesia, relief from pain. The total analgesics is comprised of prescription and non-prescription analgesics. Participants were provided with a daily diary to record the number of pills of OTC and prescription analgesics taken for endometriosis-related pain symptoms each day. The daily number of pills were standardized to a 28-day period for each interval (Baseline and On-drug Cycle 1) calculated as the sum of pills in the interval divided by the number of the days in the interval multiplied by 28. A negative change from Baseline indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to last day of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks)
Population: ITT Population consisted of all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: pills per 28-day period
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
pills per 28-day period
  Baseline | 33.8 (32.46) | 30.2 (35.09) | 74.6 (126.20)
  Change from Baseline to On-Drug Cycle | -4.96 (12.525) | -19.99 (25.132) | -12.67 (38.865)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle; Test type: Superiority; p = 0.1253, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle; Test type: Superiority; p = 0.3442, Wilcoxon Rank- Sum Test

9. Secondary Outcome: Percentage Change From Baseline in Total Analgesics Usage
Description: An analgesic was any member of the group of drugs used to achieve analgesia, relief from pain. The total analgesics is comprised of prescription and non-prescription analgesics. Participants were provided with a daily diary to record the number of pills of OTC and prescription analgesics taken for endometriosis-related pain symptoms each day. Daily number of pills were standardized to a 28-day period for each interval (Baseline and last 28-days On-drug Cycle 1) calculated as the sum of pills in the interval divided by the number of the days in the interval multiplied by 28. The percent change from baseline in the analgesic usage was determined by subtracting the baseline analgesic usage from the analgesic usage during the last nominal 28-day menstrual cycle, divided by the baseline analgesic usage, and multiplied by 100%. A negative percent change indicates improvement.
Time Frame: Baseline (28-day Baseline Menstrual Cycle) to last 28 days of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks)
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
percent change | -13.88 (64.098) | -51.96 (45.461) | -36.05 (57.129)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; On-Drug Cycle; Test type: Superiority; p = 0.0303, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; On-Drug Cycle; Test type: Superiority; p = 0.2864, Wilcoxon Rank- Sum Test

10. Secondary Outcome: Change From Baseline in BBSS Physician-Reported Scores
Description: BBSS Physician-Reported Scores included two scores: Pelvic Tenderness Score (PTS) and Induration Score (IS). PTS was graded on a scale from 0 to 3 where, 0= None; 1= Mild (minimal tenderness on palpation); 2= Moderate (extensive tenderness on palpation); 3= Severe (unable to palpate because of tenderness). IS was graded on a scale from 0 to 3 where, 0= None; 1= Mild (uterus freely mobile, induration on the cul-de-sac); 2= Moderate (thickened and indurated adnexa and cul-de-sac, restricted uterine mobility); 3= Severe (nodular adnexa and cul-de-sac, uterus frequently frozen), with higher scores indicating more severe symptoms. A negative change from Baseline indicates improvement. Data from On-drug cycle and Off-drug interval (ODI) were reported.
Time Frame: Baseline (Day 1) to last day of dosing in Cycle 1 (On-drug Cycle 1 is 18 weeks) and at the end of Off-drug Cycle 1 (Off-drug Cycle 1 is 3 weeks following On-drug Cycle 1)
Population: ITT population included all participants who were randomized and received study drug. Last observation carried forward (LOCF) approach was used to impute missing data in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
score on a scale
  PTS at Baseline (BL) | 1.9 (0.83) | 1.8 (0.77) | 1.5 (0.67)
  PTS Change from BL to LOCF Cycle 1 | -0.76 (0.903) | -0.95 (1.146) | -0.43 (0.843)
  PTS Change from BL to ODI Cycle 1: number analyzed (Participants) | 13 | 17 | 22
  PTS Change from BL to ODI Cycle 1 | -0.92 (0.954) | -0.59 (0.712) | -0.18 (1.006)
  IS at Baseline | 1.0 (1.06) | 1.1 (1.05) | 0.8 (0.83)
  IS Change from BL to LOCF Cycle 1 | -0.53 (1.007) | -0.70 (0.923) | -0.39 (0.988)
  IS Change from BL to ODI Cycle 1: number analyzed (Participants) | 13 | 17 | 22
  IS Change from BL to ODI Cycle 1 | -0.54 (0.967) | -0.59 (0.870) | -0.41 (0.796)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; PTS: LOCF Cycle 1; Test type: Superiority; p = 0.4365, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; PTS: LOCF Cycle 1; Test type: Superiority; p = 0.1302, Wilcoxon Rank- Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; PTS: ODI Cycle 1; Test type: Superiority; p = 0.3591, Wilcoxon Rank- Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; PTS: ODI Cycle 1; Test type: Superiority; p = 0.0872, Wilcoxon Rank- Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; IS: LOCF Cycle 1; Test type: Superiority; p = 0.4814, Wilcoxon Rank- Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; IS: LOCF Cycle 1; Test type: Superiority; p = 0.9162, Wilcoxon Rank- Sum Test
Statistical Analysis 7: Comparison: Placebo vs Telapristone Acetate 6 mg; IS: ODI Cycle 1; Test type: Superiority; p = 0.6607, Wilcoxon Rank- Sum Test
Statistical Analysis 8: Comparison: Placebo vs Telapristone Acetate 12 mg; IS: ODI Cycle 1; Test type: Superiority; p = 0.9527, Wilcoxon Rank- Sum Test

11. Secondary Outcome: Change From Baseline in Participant-Reported Pain Using Visual Analog Scale (VAS) Pain Score
Description: A 100-millimeter (mm) VAS was used to grade the severity of dysmenorrhea, and non-menstrual pelvic pain. The lowest value indicated the absence of pain and the highest value indicated pain as bad as it could be; a score of 1-50 was considered mild pain, 51-80 moderate pain and 81-100 severe pain. A negative change from Baseline indicates improvement. Participants were provided with a daily diary to record information about participant-reported scores for endometriosis pain.
Time Frame: as for outcome 10
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
score on a scale
  Baseline | 57.0 (27.68) | 66.6 (25.06) | 63.8 (29.14)
  Percentage change from BL to LOCF Cycle 1 | -30.11 (39.877) | -46.10 (46.871) | -17.02 (88.394)
  Percent change from BL to ODI Cycle 1: number analyzed (Participants) | 15 | 18 | 23
  Percent change from BL to ODI Cycle 1 | -29.36 (46.552) | -12.57 (52.070) | 118.34 (596.879)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; LOCF Cycle 1; Test type: Superiority; p = 0.2812, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; LOCF Cycle 1; Test type: Superiority; p = 0.5858, Wilcoxon Rank- Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; ODI Cycle 1; Test type: Superiority; p = 0.4116, Wilcoxon Rank- Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; ODI Cycle 1; Test type: Superiority; p = 0.4252, Wilcoxon Rank- Sum Test

12. Secondary Outcome: Change From Baseline in Participant-Reported Pain Using a Numerical Rating Scale (NRS)
Description: NRS is a valid and reliable clinical measure to assess pain intensity. Sex Avoidance Pain (SAP) and Endometriosis Pain (EP) were assessed using NRS-11 to measure pain based on pain ratings given by participants on the scale of 0 to 10 where, 0 represents "no pain" and 10 represents "the worst pain possible". Participants were provided with a daily diary to record information about participant-reported scores for endometriosis pain each day. Daily scores were standardized to a 28-day period for each interval (Baseline, On-drug Cycle 1 and Off-drug Cycle 1) calculated as the sum of scores in the interval divided by the number of the days in the interval multiplied by 28. A negative change from Baseline indicates improvement.
Time Frame: as for outcome 3
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: score on a scale per 28-day period
Arm/Group | Placebo | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg
Number analyzed (Participants) | 17 | 20 | 23
score on a scale per 28-day period
  SAP Baseline: number analyzed (Participants) | 8 | 14 | 19
  SAP Baseline | 67.9 (13.26) | 64.7 (15.29) | 60.6 (13.86)
  SAP Change from BL to On-Drug Cycle 1: number analyzed (Participants) | 6 | 12 | 15
  SAP Change from BL to On-Drug Cycle 1 | -2.52 (4.527) | -9.43 (14.480) | -0.53 (10.544)
  SAP Change from BL to Off-Drug Cycle 1: number analyzed (Participants) | 6 | 6 | 14
  SAP Change from BL to Off-Drug Cycle 1 | -2.21 (10.125) | -5.88 (27.822) | 3.04 (14.071)
  EP Baseline: number analyzed (Participants) | 11 | 16 | 16
  EP Baseline | 136.9 (72.48) | 136.2 (70.60) | 142.4 (70.92)
  EP Change from BL to On-Drug Cycle 1: number analyzed (Participants) | 11 | 16 | 16
  EP Change from BL to On-Drug Cycle 1 | -42.84 (39.777) | -52.05 (39.140) | -25.98 (40.954)
  EP Change from BL to Off-Drug Cycle 1: number analyzed (Participants) | 10 | 14 | 14
  EP Change from BL to Off-Drug Cycle 1 | -44.91 (43.163) | -27.06 (46.525) | -29.02 (45.496)
Statistical Analysis 1: Comparison: Placebo vs Telapristone Acetate 6 mg; SAP: On-Drug Cycle 1; Test type: Superiority; p = 0.6131, Wilcoxon Rank- Sum Test
Statistical Analysis 2: Comparison: Placebo vs Telapristone Acetate 12 mg; SAP: On-Drug Cycle 1; Test type: Superiority; p = 0.7881, Wilcoxon Rank- Sum Test
Statistical Analysis 3: Comparison: Placebo vs Telapristone Acetate 6 mg; SAP: Off-Drug Cycle 1; Test type: Superiority; p = 0.9376, Wilcoxon Rank- Sum Test
Statistical Analysis 4: Comparison: Placebo vs Telapristone Acetate 12 mg; SAP: Off-Drug Cycle 1; Test type: Superiority; p = 0.6552, Wilcoxon Rank- Sum Test
Statistical Analysis 5: Comparison: Placebo vs Telapristone Acetate 6 mg; EP: On-Drug Cycle 1; Test type: Superiority; p = 0.7143, Wilcoxon Rank- Sum Test
Statistical Analysis 6: Comparison: Placebo vs Telapristone Acetate 12 mg; EP: On-Drug Cycle 1; Test type: Superiority; p = 0.2985, Wilcoxon Rank- Sum Test
Statistical Analysis 7: Comparison: Placebo vs Telapristone Acetate 6 mg; EP: Off-Drug Cycle 1; Test type: Superiority; p = 0.3162, Wilcoxon Rank- Sum Test
Statistical Analysis 8: Comparison: Placebo vs Telapristone Acetate 12 mg; EP: Off-Drug Cycle 1; Test type: Superiority; p = 0.7503, Wilcoxon Rank- Sum Test

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately 67 weeks)
Description: AEs were reported according to the actual treatment received in Stage 2 and Stage 3.
Groups:
- Placebo (Stage 2): Following the Stage 1 no treatment baseline assessment period, placebo matching capsules, orally, once daily for 18 weeks in Stage 2. Eligible participants had the option to receive 2 additional 16-week cycles of active treatment at 12 mg/day separated by an off-drug interval (ODI) in Stage 3.
- Telapristone Acetate 6 mg (Stage 2): Following the Stage 1 no treatment baseline assessment period, telapristone acetate (Proellex®) 6 mg capsules, orally once daily for 18 weeks in Stage 2. Eligible participants had the option to receive 2 additional 16-week cycles of active treatment at 6 mg/day separated by an ODI in Stage 3.
- Telapristone Acetate 12 mg (Stage 2): Following the Stage 1 no treatment baseline assessment period, telapristone acetate (Proellex®) 12 mg capsules, orally once daily for 18 weeks. Eligible participants had the option to receive 2 additional 16-week cycles of active treatment at 12 mg/day separated by an ODI in Stage 3.
- Placebo:Telapristone Acetate 12 mg (Stage 3): Eligible participants who received placebo in Stage 2 and opted to receive up to 2 additional 16-week cycles of telapristone acetate (Proellex®) 12 mg/day in Stage 3.
- Telapristone Acetate 6 mg (Stage 3): Eligible participants who received telapristone acetate 6 mg in Stage 2 and opted to receive up to 2 additional 16-week cycles of telapristone acetate (Proellex®) 6 mg/day in Stage 3.
- Telapristone Acetate 12 mg (Stage 3): Eligible participants who received telapristone acetate 12 mg in Stage 2 and opted to receive 2 additional 16-week cycles of telapristone acetate (Proellex®) 12 mg/day in Stage 3.
Arm/Group | Placebo (Stage 2) | Telapristone Acetate 6 mg (Stage 2) | Telapristone Acetate 12 mg (Stage 2) | Placebo:Telapristone Acetate 12 mg (Stage 3) | Telapristone Acetate 6 mg (Stage 3) | Telapristone Acetate 12 mg (Stage 3)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20 | 0/23 | 0/6 | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/23 | 0/6 | 0/5 | 0/11
Other Adverse Events (participants affected / at risk) | 14/17 | 17/20 | 18/23 | 4/6 | 5/5 | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Stage 2) (N=17) | Telapristone Acetate 6 mg (Stage 2) (N=20) | Telapristone Acetate 12 mg (Stage 2) (N=23) | Placebo:Telapristone Acetate 12 mg (Stage 3) (N=6) | Telapristone Acetate 6 mg (Stage 3) (N=5) | Telapristone Acetate 12 mg (Stage 3) (N=11)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 4 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hot flush (General disorders) | 0 | 2 | 5 | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 0 | 0 | 2
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
Smear cervix abnormal (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 1 | 1
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 5 | 5 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 5 | 5 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0
Asymptomatic bacteriuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 2 | 0 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 9 | 2 | 3 | 2 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 4 | 2 | 2 | 0 | 0 | 0
Ovarian disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal infection (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vaginal odour (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Uterine haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT01728454/SAP_000.pdf
  • Study Protocol (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT01728454/Prot_001.pdf